CLINICAL TRIAL: NCT03778788
Title: A Multicentre Randomized Controlled Trial of the Effectiveness of a Lifestyle Intervention Programme Using Mobile Application vs Booklet for Adults With Metabolic Syndrome
Brief Title: a Lifestyle Intervention Programme Using Mobile Application vs Booklet for Adults With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eliza Wong, Principal Research Fellow, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HSEARS20181211005
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Metabolic Syndrome
Keywords: life style modification program; mobile application; booklet; exercise; body weight; randomized control trial; metabolic syndrome; adult
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Body Weight | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A multisite randomized controlled trial with three arms : app group, booklet and leaflet
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomizer will be used to decide the random allocation. Each eligible subject will be assigned a number generated by the computer. By using random numbers, subjects will be randomly allocated to different groups. This randomization ensure equal sample size in the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App group (Active Comparator): Participants will receive the MetS mobile application (MetS app) instalment and briefing by a research assistant (RA2) after the educational talk. They will be able view the booklet content in their own smart phone. In addition, a membership area provides individual support of self- health monitoring, goal setting for their exercise plan and exercise record.
  Interventions: Other: App group
- Booklet group (Active Comparator): The participants will additionally receive a Hong Kong version Lifestyle Intervention Programme (LIP) booklet to take home and use for 20 weeks. The major component of the LIP booklet consists of fact of metabolic syndrome, advise of diet, exercise, medication, life style and stress management.
  Interventions: Other: Booklet group
- control group (Active Comparator): Participants will be advised to maintain their usual activities. They will additionally receive a placebo health leaflet. The health leaflets are produced by Department of Health and commonly distributed to the general public. For the ethical reason, those control group participants are freely to receive the LIP booklet after completion of the study at 20 weeks.
  Interventions: Other: Booklet group; Other: control group

INTERVENTIONS:
Other: App group — Intervention group the participants will receive a Lifestyle Intervention Program (LIP) with the support of MetS mobile application (MetS app). The MetS app support include app installment and briefing by a research assistant after the educational talk. The participants can view the similar knowledge content related to metabolic syndrome in their own smart phone. In addition, a membership area provides individual support of self- health monitoring, goal setting of exercise plan and exercise record. A user guide of the MetS app will be provided to the participants to take home after the briefing.
  Arms: App group
Other: Booklet group — The participants will additionally receive a Hong Kong version LIP booklet to take home and use for 24 weeks. The major component of the LIP booklet consists of fact of metabolic syndrome, advise of diet, exercise, medication, life style and stress management.
  Arms: Booklet group; control group
Other: control group — Participants will be advised to maintain their usual activities. They will additionally receive a placebo health leaflet. The health leaflets are produced by Department of Health and commonly distributed to the general public. For the ethical reason, those control group participants are freely to receive the LIP booklet after completion of the study at 24 weeks.
  Arms: control group

SUMMARY:
The study aims to compare the effect of a lifestyle intervention programme (LIP) using mobile application (MetS app) vs using booklet for MetS adults living in the community.

DETAILED DESCRIPTION:
The study aims to compare the effect of a lifestyle intervention programme (LIP) using mobile application (MetS app) vs using booklet for MetS adults living in the community.

Methods A multi-site randomized controlled trial (RCT) with three arms, namely, MetS app group (Group A), booklet group (Group B), and control group (group C). Three hundred and sixty subjects will be recruited from six community centers and randomized into either one arm. Inclusion criteria are those MetS adult, able to use a smart phone. Group a participants will receive a 30-minute educational session and a MetS app while Group B will receive same educational session and a MetS booklet and the control group receive a placebo booklet only. The MetS app or booklet, has been well developed by the team with the support of internal grant, aims to support MetS individual's self- monitoring and record of health measures (body weight, blood pressure, waist circumference) and exercise. The primary outcomes of this study include the body weight and total physical exercise (GSLTPAQ). The secondary outcomes include cardiometabolic risk factors, cardiovascular endurance, self-efficacy for exercise (SEE) and stress level (PSS-10). Data will be collected at baseline (T1), 4 week (T2) and week 12 (T3) and week 24 (T4). SPSS and Generalized Estimating equations (GEE) model will be employed for data analysis.

Significance This study will provide empirical evidence and inform about the effective way to enhance patient's self-management of MetS, exercise sustainability that will be beneficial to clients' health.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese client who has a smart phone.
2. Adult age 18 or over
3. MetS Clients with central obesity (male >90 cm , female > 80cm ) plus two items of the followings :

   * Raised triglycerides ≥ 150 mg/dL (1.7 mmol/L) or specific treatment for this lipid abnormality
   * Reduced HDL cholesterol < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females or treatment for this lipid abnormality
   * Raised blood pressure systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension (HT)
4. Raised fasting plasma glucose (FPG) ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes (DM) -

Exclusion Criteria:

* Clients with physical, mental, visual, or cognitive impairments with regular medical follow-ups and treatment, and those who have musculoskeletal disorders or other disabling diseases that may limit the practice of walking exercise will be excluded. Client receiving prescription of medication for weight reduction will be excluded as well.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Body weight | 24 weeks
  change in body weight will be measured at the same scale in the follow up centre

SECONDARY OUTCOMES:
Total physical exercise | 24 weeks
  Total physical exercise will be quantified with a modified version of the GSLTPAQ [31-32]. The patients will be instructed to indicate the amount of exercises undertaken and rank the exercises in the order of difficulty (strenuous, moderate, or mild). The total score will be calculated. This measure has been widely used in empirical studies and shown to exhibit good Psychometric properties [31-32]
Chinese version of Self-Efficacy for Exercise (SEE-C) | 24 weeks
  The SEE-C consists of nine items, and responses are made on a 0-10 scale. The sum of the responses to all nine items yields the final composite score ranging from 0-90. The C-SE has been proved to be reliable with good psychometric properties of Cronbach's alpha coefficient 0.75 for Taiwan Chinese older adults [33-34].
Cardiovascular endurance test. | 24 weeks
  it is a three -minute step test to test the cardiovascular functional endurance after exercise across the age span and gender. A participant step on and off of a 12 inch high bench / or stair for 3 minutes. Then pulse will be taken afterward while the participant remain standing. Compare the heart rate with the table according to the age and gender to determine the fitness in a range of 7 score from excellent, good, above average, average, below average, poor and very poor . Validity of this test has been established in previous studies. [35] .
Perceived stress scale (PSS-10) | 24 weeks
  Ten self-report items measure the degree to which situations in one's life are appraised as stressful and the current levels of experienced stress in the last month. Summative scores range from 0 to 40, with a higher score indicating higher stress level. These scores have been used as outcome measures of experienced levels of stress. The psychometric properties of the Chinese version of PSS-10 were satisfactory with Cronbach's alphas >0.75 in a local study for Chinese cardiac patients. [36]
hospitalization | 24 weeks
  hospitalization frequency will be asked
app usage | 24 weeks
  MetS app usage (frequency per week) will be collected by RA by retrieving the data from the app server for the intervention group monthly.
booklet usage | 24 weeks
  Booklet usage (frequency per week) will be collected for the control group at baseline, week 4,12 and 24
Waist circumference (cm) | 24 weeks
  The Waist circumference is measured by a trained RA with a tape (cm) at the midpoint between the top of the iliac crest and the lower margin of the last rib in the standing position at the end of several consecutive natural breaths
blood pressure | 24 weeks
  Systolic and diastolic blood pressure (mmHg) is measured by a trained RA using same equipment. Data will be collected by RA
Lipid level | 24 weeks
  A drop of blood sample will be taken by using a finger stick to measure LDL cholesterol (mmol/L), and HDL cholesterol (mmol/L), and triglycerides (mmol/L). The data can be analysed immediately by using auto-analyser and the participants are asked to have 8 hours fasting. Data will be collected by RA
Fasting blood glucose | 24 weeks
  Fasting blood glucose level (mmol/L) : the participants are asked to have 8 hours fasting before blood taken. A drop of blood will be collected by finger stick by RA using same glucometer to measure the fasting blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Eliza ML Wong, Principal Investigator — HKPolyu
Locations (1):
- Wan chai Methodist Centre for the Seniors, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong EML, Tam HL, Leung AYM, Cheung ASP, Cheung KC, Leung DYP. Impacts of Educational Interventions with Support of Mobile App versus Booklet for Patients with Hypertension and Metabolic Syndrome: A Secondary Data Analysis. Int J Environ Res Public Health. 2022 Oct 2;19(19):12591. doi: 10.3390/ijerph191912591. PMID 36231891